CLINICAL TRIAL: NCT01424501
Title: Safety and Immunogenicity Study of GSK Biologicals' Candidate Tuberculosis (TB) Vaccine GSK 692342 When Administered to Adults With TB Disease
Brief Title: Safety and Immunogenicity of a Candidate Tuberculosis (TB) Vaccine in Adults With TB Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to a safety signal found at a planned interim safety review, further conduct of this safety study is not recommended hence the study was terminated.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 114886
Record Dates: First submitted 2011-08-25; First posted 2011-08-29 (Estimated); Results first posted 2017-01-24 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Tuberculosis
Keywords: Tuberculosis vaccine; HIV-negative; tuberculosis treatment
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A (Experimental): Subjects from TB-treated cohort will receive 2 doses of GSK's investigational vaccine GSK 692342.
  Interventions: Biological: GSK Biologicals' investigational TB vaccine GSK 692342
- Group B (Placebo Comparator): Subjects from TB-treated cohort will receive 2 doses of physiological Saline.
  Interventions: Biological: Placebo
- Group C (Experimental): Subjects from TB-treatment cohort will receive 2 doses of GSK's investigational vaccine GSK 692342.
  Interventions: Biological: GSK Biologicals' investigational TB vaccine GSK 692342
- Group D (Placebo Comparator): Subjects from TB-treatment cohort will receive 2 doses of physiological Saline.
  Interventions: Biological: Placebo
- Group E (Experimental): Subjects from TB-naive cohort will receive 2 doses of GSK's investigational vaccine GSK 692342.
  Interventions: Biological: GSK Biologicals' investigational TB vaccine GSK 692342
- Group F (Placebo Comparator): Subjects from TB-naive cohort will receive 2 doses of physiological Saline.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GSK Biologicals' investigational TB vaccine GSK 692342 — Intramuscular injection, 2 doses
  Arms: Group A; Group C; Group E
Biological: Placebo — Intramuscular injection, 2 doses
  Arms: Group B; Group D; Group F

SUMMARY:
This study will assess the safety and immunogenicity of GSK Biologicals' investigational tuberculosis (TB) vaccine (GSK 692342) compared to placebo when administered at 0, 1 months to human immunodeficiency virus (HIV) negative adults who have received treatment for TB disease (denoted TB-treated cohort) or are currently receiving treatment for TB disease (denoted TB-treatment cohort). For comparative purposes, subjects who have never had TB disease (denoted TB-naïve cohort) will also be enrolled.

DETAILED DESCRIPTION:
A Protocol Amendment 1, May 2012, was made following the decision to add a second country in the study (i.e. Estonia).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* A male or female between, and including, 18 and 59 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.
* Seronegative for HIV- 1 and -2 antibodies.
* No history of or current extrapulmonary tuberculosis TB. Additionally, based on medical history,
* Subjects in the TB-naive cohort must

  * have no active pulmonary disease as indicated by chest X-ray.
  * have no signs and symptoms of TB.
  * have no history of chemoprophylaxis or treatment for TB.
* Subjects in the TB-treated cohort must

  * have a history of successful treatment for pulmonary TB (completed at least 1 year prior to vaccination).
  * have no active pulmonary disease on chest X-ray.
* Subjects in the TB-treatment cohort must - have documented treatment for pulmonary TB (smear- or culture confirmed) ongoing for 2-4 months prior to vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of a registered live vaccine not foreseen by the study within 30 days preceding the first dose of study vaccine and administration of a registered inactivated vaccine within 14 days preceding the first dose of study vaccine.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Any chronic drug therapy to be continued during the study period, which in the opinion of the investigator could adversely interfere with the vaccine.
* History of previous administration of experimental TB vaccines.
* History of previous exposure to components of the investigational vaccine within 30 days preceding the first dose of study vaccine.
* Administration of any immunoglobulins, any immunotherapy and/or any blood products within the 3 months preceding the first dose of study vaccination, or planned administrations during the study period.
* Planned participation or participation in another experimental protocol during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* History of chronic alcohol and/or drug abuse.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects.
* Pregnant female, lactating female or female planning to become pregnant or discontinue contraceptive precautions during the active phase of the study (from study start till 2 months after dose 2).
* Additionally, for the TB naïve and TB treated cohorts:

  - Acute or chronic clinically relevant pulmonary, cardiovascular, hepatic or renal function abnormality as determined by physical examination or laboratory screening tests
* Additionally, for the TB treatment cohort:

  * Acute or chronic clinically relevant pulmonary, cardiovascular, hepatic or renal function abnormality as determined by physical examination or laboratory screening tests. Individuals with grade 3 levels will be excluded.
  * Failure to convert while on anti-TB treatment at the end of the second month of anti-TB therapy.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2011-11-14 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Taiwan (2):
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan Hsien

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Coccia M, Burny W, Demoitie MA, Gillard P, van den Berg RA, van der Most R. Subsequent AS01-adjuvanted vaccinations induce similar transcriptional responses in populations with different disease statuses. PLoS One. 2022 Nov 10;17(11):e0276505. doi: 10.1371/journal.pone.0276505. eCollection 2022. PMID 36355775
- [Derived] Gillard P, Yang PC, Danilovits M, Su WJ, Cheng SL, Pehme L, Bollaerts A, Jongert E, Moris P, Ofori-Anyinam O, Demoitie MA, Castro M. Safety and immunogenicity of the M72/AS01E candidate tuberculosis vaccine in adults with tuberculosis: A phase II randomised study. Tuberculosis (Edinb). 2016 Sep;100:118-127. doi: 10.1016/j.tube.2016.07.005. Epub 2016 Jul 21. PMID 27553419
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following was performed: informed consent was obtained and signed from parents or guardians of subjects, check for inclusion/exclusion criteria and contraindications/precautions, and medical history of subjects was collected. Prior to vaccination, subjects' pre-vaccination body temperature was evaluated.
Groups:
- TB Treatment GSK 692342 Group: Subjects having completed the intensive phase of treatment, i.e. 2 to 4 months post initiation of treatment, who received the GSK 692342 vaccine according to a 2-dose schedule at Months 0 and 1.
- TB Treatment Saline Group: Subjects having completed the intensive phase of treatment, i.e. 2 to 4 months post initiation of treatment who received a placebo (physiological saline) according to a 2-dose schedule at Months 0 and 1.
- TB Treated GSK 692342 Group: Subjects having successfully completed treatment for TB disease at least 1 year prior to the study, who during this study received the GSK 692342 vaccine according to a 2-dose schedule at Months 0 and 1.
- TB Treated Saline Group: Subjects having successfully completed treatment for TB disease at least 1 year prior to the study, who in this study received a placebo (physiological saline) according to a 2-dose schedule at Months 0 and 1.
- TB Naive GSK 692342 Group: Subjects unaffected by tuberculosis who received the GSK 692342 vaccine according to a 2-dose schedule at Months 0 and 1.
- TB Naive Saline Group: Subjects unaffected by tuberculosis who received a placebo (physiological saline) according to a 2-dose schedule at Months 0 and 1.
Period: Overall Study
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Started | 7 | 6 | 24 | 25 | 40 | 40
Completed | 6 | 5 | 22 | 25 | 40 | 40
Not Completed | 1 | 1 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group | Total
Number analyzed (Participants) | 7 | 6 | 24 | 25 | 40 | 40 | 142
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.9 (11.5) | 44.7 (11.8) | 44.5 (10.3) | 47 (9.8) | 33.8 (8.5) | 33.3 (9.8) | 38.7 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 13 | 7 | 16 | 21 | 60
  Male | 6 | 4 | 11 | 18 | 24 | 19 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: Asian - East Asian Heritage | 3 | 1 | 11 | 11 | 40 | 40 | 106
  Geographic ancestry: White - Caucasian/European Heritage | 4 | 5 | 13 | 14 | 0 | 0 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activities. Grade 3 redness/swelling = redness/swelling spreading beyond (>) 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with study vaccine administered, for whom data were available and who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 7 | 6 | 24 | 25 | 40 | 40
Participants
  Any Pain, Dose 1 | 6 | 1 | 21 | 2 | 38 | 5
  Grade 3 Pain, Dose 1 | 0 | 0 | 3 | 0 | 0 | 0
  Any Redness, Dose 1 | 2 | 0 | 4 | 0 | 7 | 0
  Grade 3 Redness, Dose 1 | 0 | 0 | 2 | 0 | 0 | 0
  Any Swelling, Dose 1 | 2 | 0 | 5 | 1 | 4 | 0
  Grade 3 Swelling, Dose 1 | 0 | 0 | 1 | 0 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Any Pain, Dose 2 | 5 | 1 | 19 | 1 | 36 | 6
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Grade 3 Pain, Dose 2 | 0 | 0 | 5 | 0 | 5 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Any Redness, Dose 2 | 3 | 0 | 7 | 0 | 6 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Grade 3 Redness, Dose 2 | 2 | 0 | 2 | 0 | 2 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Any Swelling, Dose 2 | 3 | 0 | 4 | 0 | 11 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Grade 3 Swelling, Dose 2 | 2 | 0 | 1 | 0 | 1 | 0
  Any Pain, Across doses | 6 | 1 | 22 | 3 | 39 | 8
  Grade 3 Pain, Across doses | 0 | 0 | 7 | 0 | 5 | 0
  Any Redness, Across doses | 3 | 0 | 8 | 0 | 10 | 0
  Grade 3 Redness, Across doses | 2 | 0 | 4 | 0 | 2 | 0
  Any Swelling, Across doses | 3 | 0 | 6 | 1 | 11 | 0
  Grade 3 Swelling, Across doses | 2 | 0 | 2 | 0 | 1 | 0

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache, malaise, myalgia and temperature [body temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of any solicited general symptom regardless of their intensity grade or relationship to vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 temperature = body temperature above (>) 39.5°C. Related = event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with study vaccine administered, for whom data were available and who had their symptoms sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 7 | 6 | 24 | 25 | 40 | 40
Participants
  Any Fatigue, Dose 1 | 1 | 2 | 14 | 6 | 19 | 8
  Grade 3 Fatigue, Dose 1 | 1 | 0 | 9 | 3 | 16 | 7
  Related Fatigue, Dose 1 | 0 | 1 | 2 | 0 | 2 | 1
  Any Gastrointestinal symptoms, Dose 1 | 0 | 0 | 4 | 2 | 5 | 5
  Grade 3 Gastrointestinal symptoms, Dose 1 | 0 | 0 | 1 | 0 | 3 | 3
  Related Gastrointestinal symptoms, Dose 1 | 0 | 0 | 2 | 0 | 0 | 0
  Any Headache, Dose 1 | 1 | 0 | 11 | 4 | 8 | 5
  Grade 3 Headache, Dose 1 | 1 | 0 | 4 | 1 | 7 | 5
  Related Headache, Dose 1 | 0 | 0 | 1 | 0 | 0 | 0
  Any Malaise, Dose 1 | 1 | 1 | 11 | 2 | 14 | 8
  Grade 3 Malaise, Dose 1 | 1 | 0 | 8 | 1 | 10 | 7
  Related Malaise, Dose 1 | 0 | 0 | 1 | 0 | 1 | 0
  Any Myalgia, Dose 1 | 2 | 0 | 13 | 4 | 24 | 7
  Grade 3 Myalgia, Dose 1 | 1 | 0 | 8 | 1 | 21 | 6
  Related Myalgia, Dose 1 | 0 | 0 | 2 | 0 | 0 | 0
  Any Temperature/(Axillary), Dose 1 | 0 | 0 | 1 | 0 | 2 | 0
  Grade 3 Temperature/(Axillary), Dose 1 | 0 | 0 | 0 | 0 | 2 | 0
  Related Temperature/(Axillary), Dose 1 | 0 | 0 | 0 | 0 | 0 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Any Fatigue, Dose 2 | 3 | 1 | 13 | 5 | 33 | 7
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Grade 3 Fatigue, Dose 2 | 3 | 0 | 11 | 0 | 30 | 7
  Related Fatigue, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Related Fatigue, Dose 2 | 0 | 0 | 2 | 0 | 3 | 0
  Any Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Any Gastrointestinal symptoms, Dose 2 | 2 | 0 | 7 | 3 | 13 | 3
  Grade 3 Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Grade 3 Gastrointestinal symptoms, Dose 2 | 0 | 0 | 5 | 0 | 11 | 3
  Related Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Related Gastrointestinal symptoms, Dose 2 | 0 | 0 | 0 | 1 | 1 | 0
  Any Headache, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Any Headache, Dose 2 | 3 | 1 | 12 | 2 | 22 | 3
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Grade 3 Headache, Dose 2 | 3 | 0 | 8 | 0 | 20 | 3
  Related Headache, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Related Headache, Dose 2 | 0 | 0 | 0 | 0 | 1 | 0
  Any Malaise, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Any Malaise, Dose 2 | 3 | 2 | 11 | 5 | 32 | 3
  Grade 3 Malaise, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Grade 3 Malaise, Dose 2 | 3 | 0 | 10 | 0 | 29 | 3
  Related Malaise, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Related Malaise, Dose 2 | 0 | 0 | 3 | 0 | 3 | 0
  Any Myalgia, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Any Myalgia, Dose 2 | 3 | 1 | 14 | 4 | 28 | 3
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Grade 3 Myalgia, Dose 2 | 3 | 0 | 13 | 1 | 27 | 3
  Related Myalgia, Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Related Myalgia, Dose 2 | 0 | 0 | 3 | 0 | 2 | 0
  Any Temperature/(Axillary), Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Any Temperature/(Axillary), Dose 2 | 4 | 1 | 9 | 0 | 16 | 0
  Grade 3 Temperature/(Axillary), Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Grade 3 Temperature/(Axillary), Dose 2 | 4 | 0 | 8 | 0 | 16 | 0
  Related Temperature/(Axillary), Dose 2: number analyzed (Participants) | 6 | 5 | 21 | 25 | 39 | 39
  Related Temperature/(Axillary), Dose 2 | 0 | 0 | 2 | 0 | 0 | 0
  Any Fatigue, Across doses | 3 | 2 | 17 | 8 | 36 | 10
  Grade 3 Fatigue, Across doses | 3 | 0 | 13 | 3 | 34 | 9
  Related Fatigue, Across doses | 0 | 1 | 4 | 0 | 5 | 1
  Any Gastrointestinal symptoms,Across doses | 2 | 0 | 10 | 4 | 16 | 6
  Grade 3 Gastrointestinal symptoms,Across doses | 0 | 0 | 6 | 0 | 13 | 4
  Related Gastrointestinal symptoms,Across doses | 0 | 0 | 2 | 1 | 1 | 0
  Any Headache, Across doses | 3 | 1 | 18 | 4 | 24 | 6
  Grade 3 Headache, Across doses | 3 | 0 | 9 | 1 | 23 | 6
  Related Headache, Across doses | 0 | 0 | 1 | 0 | 1 | 0
  Any Malaise, Across doses | 3 | 2 | 16 | 6 | 35 | 9
  Grade 3 Malaise, Across doses | 3 | 0 | 12 | 1 | 31 | 8
  Related Malaise, Across doses | 0 | 0 | 4 | 0 | 4 | 0
  Any Myalgia, Across doses | 3 | 1 | 18 | 5 | 34 | 7
  Grade 3 Myalgia, Across doses | 3 | 0 | 15 | 2 | 34 | 6
  Related Myalgia, Across doses | 0 | 0 | 5 | 0 | 2 | 0
  Any Temperature/(Axillary), Across doses | 4 | 1 | 10 | 0 | 17 | 0
  Grade 3 Temperature/(Axillary), Across doses | 4 | 0 | 8 | 0 | 17 | 0
  Related Temperature/(Axillary), Across doses | 0 | 0 | 2 | 0 | 0 | 0

3. Primary Outcome: Number of Subjects With Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: During the 30 day (Days 0-29), after vaccination
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with study vaccine administered and for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 7 | 6 | 24 | 25 | 40 | 40
Subjects | 1 | 2 | 14 | 7 | 19 | 8

4. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: Up to day 210
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 7 | 6 | 24 | 25 | 40 | 40
Subjects | 0 | 0 | 2 | 2 | 1 | 0

5. Secondary Outcome: Number of Subjects With Anti-Mycobacterium Tuberculosis Fusion Protein M72 Antibodies
Description: Cut-off values assessed were greater than or equal to (≥) 2.8, as measured by Enzyme-Linked Immunosorbent Assay (ELISA) in the sera of subjects seronegative before vaccination.
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Day 30), post-dose 2 (Days 60 and 210)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity,which included all evaluable subjects who met all eligibility criteria and complied with vaccination and blood sampling schedules,receiving a complete vaccination program or if not, they did not have blood samples taken after the interruption of the vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 7 | 4 | 21 | 25 | 38 | 39
Participants
  Anti-M72, Day 0: number analyzed (Participants) | 7 | 4 | 21 | 25 | 37 | 39
  Anti-M72, Day 0 | 0 | 0 | 0 | 0 | 1 | 2
  Anti-M72, Day 30: number analyzed (Participants) | 6 | 4 | 21 | 25 | 38 | 39
  Anti-M72, Day 30 | 5 | 0 | 19 | 0 | 26 | 2
  Anti-M72, Day 60: number analyzed (Participants) | 6 | 3 | 19 | 25 | 38 | 39
  Anti-M72, Day 60 | 6 | 0 | 18 | 0 | 37 | 3
  Anti-M72, Day 210: number analyzed (Participants) | 6 | 3 | 19 | 25 | 38 | 39
  Anti-M72, Day 210 | 6 | 0 | 18 | 0 | 38 | 1

6. Secondary Outcome: Concentrations of Anti-M72 Antibodies
Description: Concentrations are presented as geometric mean concentrations (GMCs) and expressed in ELISA units per milliliter (EU/mL).
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Day 30), post-dose 2 (Days 60 and 210)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects who met all eligibility criteria and complied with vaccination and blood sampling schedules, receiving a complete vaccination program or if not, they did not have blood samples taken after the interruption of the vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 7 | 4 | 21 | 25 | 38 | 39
EU/mL
  Anti-M72, Day 0: number analyzed (Participants) | 7 | 4 | 21 | 25 | 37 | 39
  Anti-M72, Day 0 | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.5] | 1.5 [1.4 to 1.6]
  Anti-M72, Day 30: number analyzed (Participants) | 6 | 4 | 21 | 25 | 38 | 39
  Anti-M72, Day 30 | 6.7 [2.1 to 21] | 1.4 [1.4 to 1.4] | 11.7 [6.3 to 22] | 1.4 [1.4 to 1.4] | 4.5 [3.3 to 6.2] | 1.5 [1.4 to 1.6]
  Anti-M72, Day 60: number analyzed (Participants) | 6 | 3 | 19 | 25 | 38 | 39
  Anti-M72, Day 60 | 206.6 [46.2 to 923.2] | 1.4 [1.4 to 1.4] | 226.2 [99 to 517.2] | 1.4 [1.4 to 1.4] | 248.6 [171 to 361.4] | 1.7 [1.3 to 2.3]
  Anti-M72, Day 210: number analyzed (Participants) | 6 | 3 | 19 | 25 | 38 | 39
  Anti-M72, Day 210 | 38.4 [18.9 to 77.9] | 1.4 [1.4 to 1.4] | 50.9 [27.3 to 94.8] | 1.4 [1.4 to 1.4] | 45.6 [34.2 to 60.8] | 1.4 [1.4 to 1.5]

7. Secondary Outcome: Frequency of M72-specific Cluster of Differentiation 4 (CD4+) T-cells Expressing Any Combination of the Different Immune Markers
Description: Immune markers expressed were among Interleukin-2 (IL-2), Interferon-gamma (IFN-g), Tumour necrosis factor-alpha (TNF-a) and/or CD40-ligand (CD40-L).
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD4+ T-cells/million cells
  CD4-ALL doubles, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD4-ALL doubles, Day 0 | 247 [204.5 to 333.5] | 178 [70 to 651] | 347 [196 to 523] | 549.5 [375 to 997] | 286 [173 to 471] | 352 [170 to 579]
  CD4-ALL doubles, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD4-ALL doubles, Day 7 | 997.5 [714 to 1345] | 182 [82 to 431] | 1097 [985 to 1760] | 469 [328 to 1075] | 801.5 [440 to 1492] | 265.5 [167.5 to 571.5]
  CD4-ALL doubles, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD4-ALL doubles, Day 30 | 2959 [1289 to 2989] | 730 [216 to 1244] | 2616.5 [1417 to 5614] | 466 [261.5 to 1145.5] | 1228.5 [941 to 2131] | 312.5 [202 to 726]
  CD4-ALL doubles, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD4-ALL doubles, Day 37 | 4433 [3024 to 10010] | 273 [221 to 445] | 5705.5 [2219 to 11228] | 533 [227 to 1235] | 5987.5 [3987 to 9605] | 247 [175 to 387]
  CD4-ALL doubles, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD4-ALL doubles, Day 60 | 5648 [3686 to 7957] | 241 [224 to 258] | 2072 [1083 to 4199] | 517 [352 to 1242] | 5153 [2884 to 8978] | 240 [146 to 476]
  CD4-ALL doubles, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD4-ALL doubles, Day 210 | 2922.5 [967 to 4411] | 118 [116 to 307] | 1154 [1028 to 1808] | 445 [243 to 734] | 2155 [1389 to 4160] | 254 [166 to 383]

8. Secondary Outcome: Frequency of M72-specific CD4+ T-cells Expressing at Least 2 Immune Markers Among 6
Description: Immune markers expressed were among Interleukin-2 (IL-2), Interferon-gamma (IFN-g), Tumour necrosis factor-alpha (TNF-a), CD40-ligand (CD40-L), Interleukin-17 (IL-17) and/or Interleukin-13 (IL-13).
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD4+ T-cells/million cells
  CD4-At least 2, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD4-At least 2, Day 0 | 260 [217.5 to 346.5] | 207 [96 to 687] | 364 [238 to 536] | 562.5 [402 to 1010] | 325 [240 to 512] | 365 [214 to 609]
  CD4- At least 2, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD4- At least 2, Day 7 | 1010.5 [733.5 to 1358] | 208 [95 to 457] | 1152 [1011 to 1895] | 482 [347 to 1088] | 856 [479 to 1505] | 278.5 [193.5 to 600]
  CD4- At least 2, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD4- At least 2, Day 30 | 2972 [1302 to 3002] | 765 [229 to 1301] | 2636 [1437 to 5655] | 497 [282 to 1179] | 1248.5 [954 to 2144] | 348.5 [238 to 754]
  CD4- At least 2, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD4- At least 2, Day 37 | 4446 [3037 to 10107] | 316 [234 to 458] | 5733.5 [2232 to 11281] | 565 [260 to 1262] | 6051.5 [4191 to 9679] | 277.5 [190 to 425]
  CD4- At least 2, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD4- At least 2, Day 60 | 5661 [3699 to 7976.5] | 254 [237 to 271] | 2101 [1115 to 4275] | 583 [378 to 1256] | 5185 [2897 to 9031] | 258 [160.5 to 496]
  CD4- At least 2, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD4- At least 2, Day 210 | 2948.5 [993 to 4670] | 131 [129 to 320] | 1167 [1041 to 1821] | 480 [298 to 770] | 2269 [1419 to 4173] | 299 [201.5 to 449.5]

9. Secondary Outcome: Frequency of M72-specific CD4+ T-cells Expressing Any Combination of Cytokines
Description: Immune markers (cytokines) expressed were among Interleukin-2 (IL-2), Interferon-gamma (IFN-g), Tumour necrosis factor-alpha (TNF-a) and/or CD40-ligand (CD40-L).
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD4+ T-cells/million cells
  CD40L+/IL2+/TNFa+/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2+/TNFa+/IFNg+, Day 0 | 106.5 [68 to 134] | 4 [4 to 252] | 87 [34 to 140] | 124 [74 to 186] | 60 [4 to 108] | 54 [17 to 142]
  CD40L+/IL2+/TNFa+/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2+/TNFa+/IFNg+, Day 7 | 267.5 [218.5 to 493.5] | 42 [4 to 241] | 329 [140 to 454] | 84 [25 to 154] | 87 [24 to 229] | 55.5 [4 to 132]
  CD40L+/IL2+/TNFa+/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2+/TNFa+/IFNg+, Day 30 | 1066 [261 to 1233] | 330.5 [33 to 628] | 776 [341 to 1070.5] | 71 [30.5 to 161.5] | 89.5 [37 to 287] | 47 [17 to 157]
  CD40L+/IL2+/TNFa+/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2+/TNFa+/IFNg+, Day 37 | 1186 [1084 to 1403] | 80 [44 to 158] | 897.5 [333 to 1123] | 87 [52 to 135] | 436.5 [192 to 592] | 45 [11 to 106]
  CD40L+/IL2+/TNFa+/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2+/TNFa+/IFNg+, Day 60 | 1444 [1039 to 1615.5] | 4 [4 to 4] | 417 [87 to 815] | 132 [73 to 171] | 436 [219 to 826] | 31 [4 to 130.5]
  CD40L+/IL2+/TNFa+/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2+/TNFa+/IFNg+, Day 210 | 585.5 [288 to 997] | 18 [4 to 74] | 288 [217 to 313] | 68 [38 to 157] | 201 [95 to 504] | 35.5 [18 to 89.5]
  CD40L+/IL2+/TNFa+/IFNg-, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2+/TNFa+/IFNg-, Day 0 | 12 [4 to 22] | 55 [4 to 93] | 25 [4 to 48] | 20.5 [4 to 58] | 4 [4 to 26] | 4 [4 to 33]
  CD40L+/IL2+/TNFa+/IFNg-, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2+/TNFa+/IFNg-, Day 7 | 33 [17 to 44] | 17 [4 to 45] | 44 [31 to 116] | 27 [4 to 34] | 19 [4 to 54] | 16.5 [4 to 34]
  CD40L+/IL2+/TNFa+/IFNg-, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2+/TNFa+/IFNg-, Day 30 | 204 [162 to 213] | 48 [4 to 92] | 250 [149.5 to 370.5] | 16 [4 to 43] | 279.5 [144 to 385] | 20.5 [4 to 50]
  CD40L+/IL2+/TNFa+/IFNg-, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2+/TNFa+/IFNg-, Day 37 | 436 [246 to 550] | 35 [31 to 49] | 292 [154 to 525] | 9 [4 to 43] | 558.5 [250 to 884] | 4.5 [4 to 37]
  CD40L+/IL2+/TNFa+/IFNg-, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2+/TNFa+/IFNg-, Day 60 | 654 [561.5 to 1140.5] | 28 [24 to 32] | 301 [183 to 458] | 19 [4 to 42] | 1117 [551 to 1690] | 20 [4 to 33]
  CD40L+/IL2+/TNFa+/IFNg-, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2+/TNFa+/IFNg-, Day 210 | 448 [202 to 552] | 4 [4 to 5] | 148 [116 to 209] | 18 [4 to 31] | 566 [245 to 997] | 4 [4 to 27.5]

10. Secondary Outcome: Frequency of M72-specific CD4+ T-cells Expressing Any Combination of Immune Markers
Description: as for outcome 7
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD4+ T-cells/million cells
  CD40L+/IL2+/TNFa-/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2+/TNFa-/IFNg+, Day 0 | 4 [4 to 11] | 4 [4 to 26] | 4 [4 to 23] | 17 [4 to 31] | 4 [4 to 27] | 12.5 [4 to 34]
  CD40L+/IL2+/TNFa-/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2+/TNFa-/IFNg+, Day 7 | 33 [12 to 50.5] | 4 [4 to 47] | 40 [31 to 103] | 4 [4 to 19] | 32.5 [4 to 84] | 4 [4 to 27.5]
  CD40L+/IL2+/TNFa-/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2+/TNFa-/IFNg+, Day 30 | 48 [47 to 117] | 25.5 [4 to 47] | 82.5 [39 to 116] | 4 [4 to 18.5] | 39.5 [25 to 76] | 17 [4 to 37]
  CD40L+/IL2+/TNFa-/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2+/TNFa-/IFNg+, Day 37 | 118 [89 to 307] | 4 [4 to 19] | 133.5 [42 to 242] | 4 [4 to 20] | 278 [161 to 525] | 17 [4 to 47]
  CD40L+/IL2+/TNFa-/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2+/TNFa-/IFNg+, Day 60 | 151.5 [129.5 to 246] | 32 [4 to 60] | 75 [44 to 236] | 4 [4 to 18] | 269 [128 to 500] | 4 [4 to 28.5]
  CD40L+/IL2+/TNFa-/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2+/TNFa-/IFNg+, Day 210 | 112.5 [31 to 218] | 18 [4 to 60] | 47 [24 to 95] | 4 [4 to 29] | 126 [61 to 296] | 10.5 [4 to 40]
  CD40L+/IL2+/TNFa-/IFNg-, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2+/TNFa-/IFNg-, Day 0 | 11.5 [4 to 41] | 4 [4 to 17] | 14 [4 to 22] | 17.5 [4 to 45] | 19.5 [4 to 37] | 4 [4 to 24]
  CD40L+/IL2+/TNFa-/IFNg-, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2+/TNFa-/IFNg-, Day 7 | 45.5 [4 to 88] | 4 [4 to 17] | 43 [17 to 75] | 4 [4 to 46] | 44.5 [4 to 69] | 5 [4 to 49.5]
  CD40L+/IL2+/TNFa-/IFNg-, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2+/TNFa-/IFNg-, Day 30 | 102 [32 to 201] | 84.5 [33 to 136] | 150.5 [69 to 253.5] | 25 [4 to 53] | 300 [202 to 519] | 18 [4 to 49]
  CD40L+/IL2+/TNFa-/IFNg-, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2+/TNFa-/IFNg-, Day 37 | 263 [94 to 305] | 20 [4 to 65] | 182 [67 to 393] | 4 [4 to 29] | 732 [498 to 946] | 4 [4 to 16]
  CD40L+/IL2+/TNFa-/IFNg-, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2+/TNFa-/IFNg-, Day 60 | 381.5 [223.5 to 561.5] | 46.5 [32 to 61] | 171 [84 to 514] | 4 [4 to 38] | 939 [534 to 1537] | 17.5 [4 to 30]
  CD40L+/IL2+/TNFa-/IFNg-, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2+/TNFa-/IFNg-, Day 210 | 166.5 [66 to 380] | 18 [4 to 31] | 126 [101 to 148] | 17 [4 to 32] | 453 [281 to 768] | 11 [4 to 37]

11. Secondary Outcome: Frequency of CD4+ T-cells M72-specific Expressing Any Combination of Cytokines
Description: as for outcome 9
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD4+ T-cells/million cells
  CD40L+/IL2-/TNFa+/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2-/TNFa+/IFNg+, Day 0 | 67 [47 to 74.5] | 55 [4 to 161] | 61 [19 to 218] | 188.5 [66 to 272] | 48.5 [17 to 101] | 44.5 [19 to 164]
  CD40L+/IL2-/TNFa+/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2-/TNFa+/IFNg+, Day 7 | 270.5 [224 to 408.5] | 4 [4 to 73] | 389 [207 to 735] | 151 [79 to 278] | 232 [46 to 491] | 43 [10.5 to 148.5]
  CD40L+/IL2-/TNFa+/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2-/TNFa+/IFNg+, Day 30 | 563 [541 to 1023] | 115 [4 to 226] | 902 [397.5 to 2177] | 132.5 [54.5 to 398] | 156.5 [76 to 481] | 71.5 [18 to 221]
  CD40L+/IL2-/TNFa+/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2-/TNFa+/IFNg+, Day 37 | 1236 [886 to 3361] | 4 [4 to 111] | 1828 [462 to 3273] | 253 [45 to 463] | 738.5 [422 to 1663] | 46.5 [17 to 114]
  CD40L+/IL2-/TNFa+/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2-/TNFa+/IFNg+, Day 60 | 2219.5 [1183 to 3234] | 24.5 [4 to 45] | 608 [361 to 1433] | 149.5 [97 to 340] | 560 [192 to 1563] | 55.5 [25.5 to 150]
  CD40L+/IL2-/TNFa+/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2-/TNFa+/IFNg+, Day 210 | 869 [202 to 1422] | 32 [4 to 33] | 439 [218 to 620] | 174 [46 to 248] | 301 [137 to 602] | 22 [4 to 137]
  CD40L+/IL2-/TNFa+/IFNg-, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2-/TNFa+/IFNg-, Day 0 | 10 [4 to 20.5] | 20 [4 to 73] | 8 [4 to 38] | 18 [4 to 43] | 9.5 [4 to 47] | 20 [4 to 52]
  CD40L+/IL2-/TNFa+/IFNg-, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2-/TNFa+/IFNg-, Day 7 | 34 [18 to 40.5] | 17 [4 to 47] | 58 [24 to 74] | 4 [4 to 31] | 40.5 [17 to 98] | 4 [4 to 41]
  CD40L+/IL2-/TNFa+/IFNg-, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2-/TNFa+/IFNg-, Day 30 | 132 [45 to 150] | 25.5 [4 to 47] | 152.5 [79 to 215] | 25.5 [4 to 52.5] | 125.5 [71 to 216] | 17 [4 to 28]
  CD40L+/IL2-/TNFa+/IFNg-, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2-/TNFa+/IFNg-, Day 37 | 276 [117 to 889] | 37 [4 to 87] | 375.5 [230 to 805] | 40 [4 to 84] | 915 [471 to 1575] | 18 [4 to 38]
  CD40L+/IL2-/TNFa+/IFNg-, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2-/TNFa+/IFNg-, Day 60 | 359.5 [255 to 556.5] | 62.5 [4 to 121] | 176 [75 to 327] | 26 [4 to 65] | 792 [421 to 1060] | 4 [4 to 38.5]
  CD40L+/IL2-/TNFa+/IFNg-, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2-/TNFa+/IFNg-, Day 210 | 167 [75 to 191] | 19 [4 to 35] | 77 [23 to 134] | 4 [4 to 40] | 272 [142 to 358] | 18 [4 to 34.5]

12. Secondary Outcome: Frequency of CD4+ T-cells M72-specific Expressing Any Combination of Immune Markers
Description: as for outcome 7
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD4+ T-cells/million cells
  CD40L+/IL2-/TNFa-/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2-/TNFa-/IFNg+, Day 0 | 10.5 [4 to 40] | 17 [4 to 20] | 25 [6 to 61] | 43 [4 to 80] | 27.5 [4 to 54] | 12 [4 to 60]
  CD40L+/IL2-/TNFa-/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2-/TNFa-/IFNg+, Day 7 | 113.5 [62.5 to 155.5] | 4 [4 to 31] | 227 [65 to 469] | 22 [4 to 71] | 163 [100 to 239] | 29.5 [4 to 54]
  CD40L+/IL2-/TNFa-/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2-/TNFa-/IFNg+, Day 30 | 71 [60 to 75] | 41 [32 to 50] | 124.5 [64.5 to 284] | 13.5 [4 to 65] | 86.5 [27 to 154] | 30 [4 to 59]
  CD40L+/IL2-/TNFa-/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2-/TNFa-/IFNg+, Day 37 | 406 [406 to 1923] | 5 [4 to 31] | 649 [245 to 1982] | 17 [4 to 72] | 1355.5 [917 to 2882] | 19 [4 to 58]
  CD40L+/IL2-/TNFa-/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2-/TNFa-/IFNg+, Day 60 | 213 [75 to 378.5] | 17.5 [4 to 31] | 147 [58 to 339] | 20.5 [4 to 46] | 399 [135 to 664] | 4 [4 to 35.5]
  CD40L+/IL2-/TNFa-/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2-/TNFa-/IFNg+, Day 210 | 129 [18 to 304] | 4 [4 to 73] | 57 [37 to 115] | 32 [4 to 62] | 107 [65 to 180] | 30.5 [5 to 48]
  CD40L+/IL2-/TNFa-/IFNg-, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2-/TNFa-/IFNg-, Day 0 | 4 [4 to 98.5] | 103 [4 to 244] | 19 [4 to 41] | 10.5 [4 to 73] | 4 [4 to 29] | 4 [4 to 32]
  CD40L+/IL2-/TNFa-/IFNg-, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2-/TNFa-/IFNg-, Day 7 | 4 [4 to 10.5] | 4 [4 to 506] | 14 [4 to 83] | 4 [4 to 23] | 19 [4 to 171] | 4 [4 to 41.5]
  CD40L+/IL2-/TNFa-/IFNg-, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2-/TNFa-/IFNg-, Day 30 | 4 [4 to 18] | 1375.5 [4 to 2747] | 208 [11 to 689] | 4 [4 to 37] | 342 [133 to 769] | 4 [4 to 136]
  CD40L+/IL2-/TNFa-/IFNg-, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2-/TNFa-/IFNg-, Day 37 | 937 [17 to 1644] | 213 [20 to 373] | 1544 [787 to 2630] | 18 [4 to 200] | 3575.5 [2450 to 6212] | 4 [4 to 32]
  CD40L+/IL2-/TNFa-/IFNg-, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2-/TNFa-/IFNg-, Day 60 | 4 [4 to 373.5] | 4 [4 to 4] | 168 [4 to 727] | 4 [4 to 104] | 1426 [653 to 2820] | 4 [4 to 89]
  CD40L+/IL2-/TNFa-/IFNg-, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2-/TNFa-/IFNg-, Day 210 | 10.5 [4 to 712] | 4 [4 to 4] | 296 [13 to 743] | 45 [4 to 233] | 497 [34 to 900] | 4 [4 to 89.5]

13. Secondary Outcome: Frequency of M72-specific CD4+ T-cells Expressing Cytokines in Any Combination
Description: as for outcome 9
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD4+ T-cells/million cells
  CD40L-/IL2+/TNFa+/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L-/IL2+/TNFa+/IFNg+, Day 0 | 4 [4 to 4] | 4 [4 to 26] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L-/IL2+/TNFa+/IFNg+, Day 7 | 4 [4 to 68] | 4 [4 to 17] | 19 [4 to 74] | 4 [4 to 18] | 4 [4 to 26] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L-/IL2+/TNFa+/IFNg+, Day 30 | 4 [4 to 41] | 26 [4 to 48] | 35 [4 to 85] | 4 [4 to 10.5] | 4 [4 to 25] | 4 [4 to 19]
  CD40L-/IL2+/TNFa+/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L-/IL2+/TNFa+/IFNg+, Day 37 | 89 [46 to 93] | 4 [4 to 4] | 64.5 [17 to 148] | 4 [4 to 4] | 32.5 [4 to 66] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L-/IL2+/TNFa+/IFNg+, Day 60 | 39.5 [17.5 to 62.5] | 4 [4 to 4] | 4 [4 to 60] | 4 [4 to 4] | 19 [4 to 33] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L-/IL2+/TNFa+/IFNg+, Day 210 | 19 [4 to 32] | 4 [4 to 4] | 4 [4 to 19] | 4 [4 to 4] | 4 [4 to 31] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg-, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L-/IL2+/TNFa+/IFNg-, Day 0 | 4 [4 to 11] | 4 [4 to 4] | 4 [4 to 20] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg-, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L-/IL2+/TNFa+/IFNg-, Day 7 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg-, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L-/IL2+/TNFa+/IFNg-, Day 30 | 17 [4 to 17] | 4 [4 to 4] | 19.5 [4 to 54.5] | 4 [4 to 17.5] | 17.5 [4 to 33] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg-, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L-/IL2+/TNFa+/IFNg-, Day 37 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 24] | 4 [4 to 4] | 34 [8 to 67] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg-, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L-/IL2+/TNFa+/IFNg-, Day 60 | 21 [10.5 to 55.5] | 4 [4 to 4] | 4 [4 to 19] | 4 [4 to 4] | 45 [16 to 79] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg-, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L-/IL2+/TNFa+/IFNg-, Day 210 | 4 [4 to 21] | 17 [4 to 18] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 34] | 4 [4 to 10.5]

14. Secondary Outcome: Frequency of M72-specific CD4+ T-cells Expressing Immune Markers in Any Combination
Description: as for outcome 7
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD4+ T-cells/million cells
  CD40L-/IL2+/TNFa-/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L-/IL2+/TNFa-/IFNg+, Day 0 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa-/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L-/IL2+/TNFa-/IFNg+, Day 7 | 4 [4 to 16.5] | 4 [4 to 4] | 17 [4 to 18] | 4 [4 to 4] | 4 [4 to 19] | 4 [4 to 4]
  CD40L-/IL2+/TNFa-/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L-/IL2+/TNFa-/IFNg+, Day 30 | 4 [4 to 4] | 4 [4 to 4] | 11 [4 to 23.5] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa-/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L-/IL2+/TNFa-/IFNg+, Day 37 | 17 [17 to 32] | 4 [4 to 4] | 17 [4 to 24] | 4 [4 to 4] | 19.5 [4 to 61] | 4 [4 to 4]
  CD40L-/IL2+/TNFa-/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L-/IL2+/TNFa-/IFNg+, Day 60 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 20] | 4 [4 to 4] | 4 [4 to 22] | 4 [4 to 4]
  CD40L-/IL2+/TNFa-/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L-/IL2+/TNFa-/IFNg+, Day 210 | 4 [4 to 24] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa-/IFNg-, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L-/IL2+/TNFa-/IFNg-, Day 0 | 4 [4 to 10.5] | 4 [4 to 20] | 4 [4 to 23] | 4 [4 to 18] | 4 [4 to 4] | 4 [4 to 21]
  CD40L-/IL2+/TNFa-/IFNg-, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L-/IL2+/TNFa-/IFNg-, Day 7 | 4 [4 to 18] | 4 [4 to 17] | 4 [4 to 17] | 17 [4 to 30] | 18.5 [4 to 26] | 4 [4 to 12]
  CD40L-/IL2+/TNFa-/IFNg-, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L-/IL2+/TNFa-/IFNg-, Day 30 | 30 [19 to 32] | 4 [4 to 4] | 21 [6.5 to 44.5] | 4 [4 to 19] | 18 [4 to 32] | 4 [4 to 20]
  CD40L-/IL2+/TNFa-/IFNg-, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L-/IL2+/TNFa-/IFNg-, Day 37 | 4 [4 to 4] | 4 [4 to 4] | 27.5 [17 to 45] | 4 [4 to 5] | 40.5 [19 to 82] | 4 [4 to 20]
  CD40L-/IL2+/TNFa-/IFNg-, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L-/IL2+/TNFa-/IFNg-, Day 60 | 11 [4.5 to 28.5] | 17.5 [4 to 31] | 4 [4 to 20] | 11 [4 to 23] | 49 [20 to 70] | 4 [4 to 18]
  CD40L-/IL2+/TNFa-/IFNg-, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L-/IL2+/TNFa-/IFNg-, Day 210 | 17.5 [4 to 59] | 4 [4 to 32] | 4 [4 to 17] | 4 [4 to 26] | 25 [8 to 44] | 4 [4 to 19.5]

15. Secondary Outcome: Frequency of CD4+ T-cells M72-specific Expressing Cytokines in Any Combination
Description: as for outcome 9
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD4+ T-cells/million cells
  CD40L-/IL2-/TNFa+/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L-/IL2-/TNFa+/IFNg+, Day 0 | 10.5 [4 to 25] | 4 [4 to 4] | 24 [4 to 59] | 13.5 [4 to 136] | 17.5 [4 to 32] | 4 [4 to 57]
  CD40L-/IL2-/TNFa+/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L-/IL2-/TNFa+/IFNg+, Day 7 | 53.5 [34.5 to 87.5] | 4 [4 to 17] | 102 [40 to 230] | 18 [4 to 234] | 53 [17 to 246] | 4 [4 to 53]
  CD40L-/IL2-/TNFa+/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L-/IL2-/TNFa+/IFNg+, Day 30 | 76 [4 to 117] | 26 [4 to 48] | 112 [21.5 to 212] | 44 [10.5 to 334.5] | 42 [4 to 89] | 20 [4 to 46]
  CD40L-/IL2-/TNFa+/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L-/IL2-/TNFa+/IFNg+, Day 37 | 246 [116 to 288] | 34 [4 to 65] | 212.5 [94 to 698] | 50 [5 to 361] | 185.5 [61 to 463] | 4 [4 to 33]
  CD40L-/IL2-/TNFa+/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L-/IL2-/TNFa+/IFNg+, Day 60 | 162.5 [76 to 214] | 14 [4 to 24] | 34 [19 to 338] | 46 [4 to 534] | 69 [32 to 277] | 18.5 [4 to 45.5]
  CD40L-/IL2-/TNFa+/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L-/IL2-/TNFa+/IFNg+, Day 210 | 19.5 [4 to 156] | 4 [4 to 18] | 30 [18 to 112] | 29 [4 to 169] | 46 [4 to 77] | 11.5 [4 to 38]
  CD40L-/IL2-/TNFa+/IFNg-, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L-/IL2-/TNFa+/IFNg-, Day 0 | 11.5 [5 to 31] | 18 [18 to 29] | 20 [4 to 55] | 4 [4 to 41] | 8 [4 to 38] | 22.5 [4 to 68]
  CD40L-/IL2-/TNFa+/IFNg-, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L-/IL2-/TNFa+/IFNg-, Day 7 | 25.5 [11 to 38] | 17 [4 to 45] | 19 [4 to 75] | 17 [4 to 32] | 26 [4 to 57] | 28.5 [4 to 81.5]
  CD40L-/IL2-/TNFa+/IFNg-, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L-/IL2-/TNFa+/IFNg-, Day 30 | 21 [6 to 26] | 4 [4 to 4] | 51.5 [15 to 101] | 32.5 [4.5 to 67] | 8 [4 to 61] | 12.5 [4 to 31]
  CD40L-/IL2-/TNFa+/IFNg-, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L-/IL2-/TNFa+/IFNg-, Day 37 | 46 [31 to 153] | 66 [31 to 117] | 87 [31 to 256] | 11 [4 to 119] | 309 [137 to 532] | 7.5 [4 to 26]
  CD40L-/IL2-/TNFa+/IFNg-, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L-/IL2-/TNFa+/IFNg-, Day 60 | 67 [57.5 to 108] | 50 [40 to 60] | 23 [4 to 104] | 36 [4 to 59] | 88 [35 to 225] | 22 [4 to 44]
  CD40L-/IL2-/TNFa+/IFNg-, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L-/IL2-/TNFa+/IFNg-, Day 210 | 4 [4 to 60] | 4 [4 to 4] | 5 [4 to 57] | 23 [4 to 54] | 24 [4 to 76] | 4 [4 to 34.5]

16. Secondary Outcome: Frequency of CD4+ T-cells M72-specific Expressing Immune Markers in Any Combination
Description: as for outcome 7
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD4+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD4+ T-cells/million cells
  CD40L-/IL2-/TNFa-/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L-/IL2-/TNFa-/IFNg+, Day 0 | 17.5 [4 to 52.5] | 20 [4 to 61] | 47 [4 to 64] | 51 [4 to 99] | 70 [38 to 157] | 14.5 [4 to 85]
  CD40L-/IL2-/TNFa-/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L-/IL2-/TNFa-/IFNg+, Day 7 | 69.5 [17.5 to 114] | 4 [4 to 83] | 59 [12 to 363] | 46 [6 to 482] | 78 [32 to 248] | 25.5 [4 to 76]
  CD40L-/IL2-/TNFa-/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L-/IL2-/TNFa-/IFNg+, Day 30 | 45 [45 to 61] | 4 [4 to 4] | 52 [4 to 201.5] | 33.5 [4 to 270] | 47 [4 to 138] | 26.5 [4 to 132]
  CD40L-/IL2-/TNFa-/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L-/IL2-/TNFa-/IFNg+, Day 37 | 191 [89 to 408] | 34 [31 to 97] | 273 [131 to 720] | 27 [4 to 261] | 495.5 [267 to 1466] | 19 [4 to 86]
  CD40L-/IL2-/TNFa-/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L-/IL2-/TNFa-/IFNg+, Day 60 | 14.5 [4 to 48.5] | 4 [4 to 4] | 32 [4 to 267] | 51.5 [17 to 144] | 129 [40 to 276] | 19.5 [4 to 84]
  CD40L-/IL2-/TNFa-/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L-/IL2-/TNFa-/IFNg+, Day 210 | 53.5 [31 to 117] | 4 [4 to 60] | 30 [4 to 85] | 34 [4 to 92] | 31 [4 to 126] | 55 [32.5 to 115]

17. Secondary Outcome: Frequency of M72-specific Cluster of Differentiation 8 (CD8+) T-cells Expressing at Least 2 Immune Markers
Description: as for outcome 7
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD8+ T-cells/million cells
  CD8-All Doubles, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD8-All Doubles, Day 0 | 93 [63.5 to 269] | 44 [44 to 135] | 99 [75 to 159] | 110.5 [59 to 326] | 73 [44 to 144] | 69.5 [44 to 132]
  CD8-All Doubles, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD8-All Doubles, Day 7 | 94.5 [80.5 to 141] | 72 [45 to 77] | 222 [146 to 329] | 62 [44 to 324] | 74.5 [44 to 144] | 92.5 [53 to 191]
  CD8-All Doubles, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD8-All Doubles, Day 30 | 44 [44 to 64] | 81.5 [44 to 119] | 243 [101 to 385] | 153.5 [75.5 to 1064] | 80 [44 to 150] | 77.5 [59 to 172]
  CD8-All Doubles, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD8-All Doubles, Day 37 | 126 [118 to 134] | 76 [44 to 93] | 347 [97 to 604] | 108 [59 to 295] | 72.5 [57 to 149] | 75.5 [44 to 140]
  CD8-All Doubles, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD8-All Doubles, Day 60 | 85.5 [55.5 to 233] | 118 [69 to 167] | 189 [60 to 367] | 161 [84 to 491] | 96 [44 to 245] | 71 [44 to 157.5]
  CD8-All Doubles, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD8-All Doubles, Day 210 | 347.5 [170 to 572] | 78 [44 to 91] | 259 [61 to 312] | 119 [44 to 390] | 110 [69 to 248] | 71.5 [49.5 to 233]

18. Secondary Outcome: Frequency of M72-specific CD8+ T-cells Expressing at Least 2 Immune Markers Among 6
Description: as for outcome 8
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD8+ T-cells/million cells
  CD8-At least 2, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD8-At least 2, Day 0 | 106 [76.5 to 282] | 57 [57 to 148] | 143 [88 to 172] | 151.5 [81 to 339] | 96 [57 to 157] | 85.5 [57 to 169]
  CD8- At least 2, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD8- At least 2, Day 7 | 107.5 [93.5 to 154] | 85 [58 to 90] | 245 [159 to 369] | 75 [57 to 337] | 116 [71 to 158] | 124 [88 to 232]
  CD8- At least 2, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD8- At least 2, Day 30 | 57 [57 to 77] | 109 [86 to 132] | 256 [114 to 410.5] | 166.5 [88.5 to 1077] | 96 [73 to 163] | 106.5 [77 to 198]
  CD8- At least 2, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD8- At least 2, Day 37 | 139 [131 to 147] | 89 [57 to 106] | 362 [110 to 617] | 121 [72 to 308] | 85.5 [70 to 162] | 103.5 [58 to 161]
  CD8- At least 2, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD8- At least 2, Day 60 | 98.5 [68.5 to 246] | 131 [82 to 180] | 202 [89 to 380] | 174 [97 to 504] | 111 [76 to 270] | 106.5 [57 to 191]
  CD8- At least 2, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD8- At least 2, Day 210 | 403.5 [183 to 585] | 91 [57 to 151] | 272 [74 to 379] | 133 [76 to 403] | 137 [83 to 291] | 124.5 [81.5 to 292]

19. Secondary Outcome: Frequency of M72-specific CD8+ T-cells Expressing Any Combination of Immune Markers
Description: as for outcome 7
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD8+ T-cells/million cells
  CD40L+/IL2+/TNFa+/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2+/TNFa+/IFNg+, Day 0 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa+/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2+/TNFa+/IFNg+, Day 7 | 4 [4 to 14] | 4 [4 to 4] | 4 [4 to 62] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa+/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2+/TNFa+/IFNg+, Day 30 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 25] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa+/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2+/TNFa+/IFNg+, Day 37 | 4 [4 to 41] | 4 [4 to 4] | 4 [4 to 48] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa+/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2+/TNFa+/IFNg+, Day 60 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa+/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2+/TNFa+/IFNg+, Day 210 | 58 [4 to 99] | 4 [4 to 38] | 4 [4 to 4] | 4 [4 to 33] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa+/IFNg-, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2+/TNFa+/IFNg-, Day 0 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa+/IFNg-, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2+/TNFa+/IFNg-, Day 7 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa+/IFNg-, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2+/TNFa+/IFNg-, Day 30 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa+/IFNg-, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2+/TNFa+/IFNg-, Day 37 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa+/IFNg-, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2+/TNFa+/IFNg-, Day 60 | 4 [4 to 19] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa+/IFNg-, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2+/TNFa+/IFNg-, Day 210 | 35 [4 to 46] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 25] | 4 [4 to 4]

20. Secondary Outcome: Frequency of M72-specific CD8+ T-cells Expressing Any Combination of Cytokines
Description: as for outcome 9
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD8+ T-cells/million cells
  CD40L+/IL2+/TNFa-/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2+/TNFa-/IFNg+, Day 0 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa-/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2+/TNFa-/IFNg+, Day 7 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa-/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2+/TNFa-/IFNg+, Day 30 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa-/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2+/TNFa-/IFNg+, Day 37 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa-/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2+/TNFa-/IFNg+, Day 60 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa-/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2+/TNFa-/IFNg+, Day 210 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa-/IFNg-, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2+/TNFa-/IFNg-, Day 0 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa-/IFNg-, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2+/TNFa-/IFNg-, Day 7 | 4 [4 to 4] | 4 [4 to 32] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa-/IFNg-, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2+/TNFa-/IFNg-, Day 30 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa-/IFNg-, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2+/TNFa-/IFNg-, Day 37 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa-/IFNg-, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2+/TNFa-/IFNg-, Day 60 | 4 [4 to 4] | 14 [4 to 24] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2+/TNFa-/IFNg-, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2+/TNFa-/IFNg-, Day 210 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]

21. Secondary Outcome: Frequency of CD8+ T-cells M72-specific Expressing Any Combination of Immune Markers
Description: as for outcome 7
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD8+ T-cells/million cells
  CD40L+/IL2-/TNFa+/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2-/TNFa+/IFNg+, Day 0 | 4 [4 to 33.5] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 23] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2-/TNFa+/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2-/TNFa+/IFNg+, Day 7 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 55] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2-/TNFa+/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2-/TNFa+/IFNg+, Day 30 | 4 [4 to 4] | 4 [4 to 4] | 36.5 [4 to 84] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2-/TNFa+/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2-/TNFa+/IFNg+, Day 37 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 168] | 4 [4 to 21] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2-/TNFa+/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2-/TNFa+/IFNg+, Day 60 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 42] | 4 [4 to 24] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2-/TNFa+/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2-/TNFa+/IFNg+, Day 210 | 4 [4 to 13] | 4 [4 to 51] | 4 [4 to 56] | 4 [4 to 4] | 4 [4 to 21] | 4 [4 to 4]
  CD40L+/IL2-/TNFa+/IFNg-, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2-/TNFa+/IFNg-, Day 0 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2-/TNFa+/IFNg-, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2-/TNFa+/IFNg-, Day 7 | 4 [4 to 4] | 4 [4 to 37] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2-/TNFa+/IFNg-, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2-/TNFa+/IFNg-, Day 30 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 17] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2-/TNFa+/IFNg-, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2-/TNFa+/IFNg-, Day 37 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2-/TNFa+/IFNg-, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2-/TNFa+/IFNg-, Day 60 | 4 [4 to 21] | 24.5 [4 to 45] | 4 [4 to 20] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L+/IL2-/TNFa+/IFNg-, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2-/TNFa+/IFNg-, Day 210 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 21] | 4 [4 to 4] | 4 [4 to 19] | 4 [4 to 9]

22. Secondary Outcome: Frequency of CD8+ T-cells M72-specific Expressing Any Combination of Cytokines
Description: as for outcome 9
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD8+ T-cells/million cells
  CD40L+/IL2-/TNFa-/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2-/TNFa-/IFNg+, Day 0 | 4 [4 to 23.5] | 4 [4 to 26] | 4 [4 to 5] | 4 [4 to 4] | 4 [4 to 26] | 4 [4 to 18]
  CD40L+/IL2-/TNFa-/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2-/TNFa-/IFNg+, Day 7 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 54] | 4 [4 to 22] | 4 [4 to 24] | 4 [4 to 4.5]
  CD40L+/IL2-/TNFa-/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2-/TNFa-/IFNg+, Day 30 | 4 [4 to 4] | 41.5 [4 to 79] | 4 [4 to 4] | 4 [4 to 28.5] | 4 [4 to 25] | 4 [4 to 31]
  CD40L+/IL2-/TNFa-/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2-/TNFa-/IFNg+, Day 37 | 4 [4 to 4] | 4 [4 to 36] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 21] | 4 [4 to 23]
  CD40L+/IL2-/TNFa-/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2-/TNFa-/IFNg+, Day 60 | 4 [4 to 21] | 16.5 [4 to 29] | 4 [4 to 4] | 14.5 [4 to 46] | 4 [4 to 76] | 4 [4 to 14.5]
  CD40L+/IL2-/TNFa-/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2-/TNFa-/IFNg+, Day 210 | 19.5 [4 to 88] | 4 [4 to 4] | 4 [4 to 35] | 4 [4 to 4] | 4 [4 to 29] | 4 [4 to 34.5]
  CD40L+/IL2-/TNFa-/IFNg-, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L+/IL2-/TNFa-/IFNg-, Day 0 | 97.5 [4 to 412] | 143 [4 to 178] | 29 [4 to 203] | 4 [4 to 139] | 7.5 [4 to 130] | 25 [4 to 222]
  CD40L+/IL2-/TNFa-/IFNg-, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L+/IL2-/TNFa-/IFNg-, Day 7 | 33.5 [4 to 68] | 110 [93 to 390] | 4 [4 to 4] | 4 [4 to 413] | 4 [4 to 183] | 26 [4 to 164]
  CD40L+/IL2-/TNFa-/IFNg-, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L+/IL2-/TNFa-/IFNg-, Day 30 | 73 [4 to 113] | 161 [83 to 239] | 4 [4 to 23] | 4 [4 to 78.5] | 4 [4 to 71] | 99.5 [4 to 288]
  CD40L+/IL2-/TNFa-/IFNg-, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L+/IL2-/TNFa-/IFNg-, Day 37 | 4 [4 to 203] | 4 [4 to 216] | 4 [4 to 293] | 43 [4 to 125] | 4 [4 to 127] | 13.5 [4 to 213]
  CD40L+/IL2-/TNFa-/IFNg-, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L+/IL2-/TNFa-/IFNg-, Day 60 | 18.5 [4 to 163.5] | 44.5 [4 to 85] | 101 [4 to 345] | 85 [4 to 270] | 61 [4 to 153] | 36.5 [4 to 214]
  CD40L+/IL2-/TNFa-/IFNg-, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L+/IL2-/TNFa-/IFNg-, Day 210 | 53 [15 to 92] | 122 [4 to 202] | 333 [4 to 583] | 121 [4 to 249] | 22 [4 to 311] | 33.5 [4 to 302.5]

23. Secondary Outcome: Frequency of M72-specific CD8+ T-cells Expressing Cytokines in Any Combination
Description: as for outcome 9
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD8+ T-cells/million cells
  CD40L-/IL2+/TNFa+/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L-/IL2+/TNFa+/IFNg+, Day 0 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L-/IL2+/TNFa+/IFNg+, Day 7 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L-/IL2+/TNFa+/IFNg+, Day 30 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L-/IL2+/TNFa+/IFNg+, Day 37 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L-/IL2+/TNFa+/IFNg+, Day 60 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L-/IL2+/TNFa+/IFNg+, Day 210 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg-, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L-/IL2+/TNFa+/IFNg-, Day 0 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg-, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L-/IL2+/TNFa+/IFNg-, Day 7 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg-, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L-/IL2+/TNFa+/IFNg-, Day 30 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg-, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L-/IL2+/TNFa+/IFNg-, Day 37 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg-, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L-/IL2+/TNFa+/IFNg-, Day 60 | 4 [4 to 15.5] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa+/IFNg-, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L-/IL2+/TNFa+/IFNg-, Day 210 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]

24. Secondary Outcome: Frequency of M72-specific CD8+ T-cells Expressing Immune Markers in Any Combination
Description: as for outcome 7
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD8+ T-cells/million cells
  CD40L-/IL2+/TNFa-/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L-/IL2+/TNFa-/IFNg+, Day 0 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa-/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L-/IL2+/TNFa-/IFNg+, Day 7 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa-/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L-/IL2+/TNFa-/IFNg+, Day 30 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa-/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L-/IL2+/TNFa-/IFNg+, Day 37 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa-/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L-/IL2+/TNFa-/IFNg+, Day 60 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa-/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L-/IL2+/TNFa-/IFNg+, Day 210 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4]
  CD40L-/IL2+/TNFa-/IFNg-, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L-/IL2+/TNFa-/IFNg-, Day 0 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 41] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 5]
  CD40L-/IL2+/TNFa-/IFNg-, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L-/IL2+/TNFa-/IFNg-, Day 7 | 4 [4 to 4] | 4 [4 to 37] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 20] | 4 [4 to 23.5]
  CD40L-/IL2+/TNFa-/IFNg-, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L-/IL2+/TNFa-/IFNg-, Day 30 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 32] | 4 [4 to 4] | 4 [4 to 19] | 4 [4 to 4]
  CD40L-/IL2+/TNFa-/IFNg-, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L-/IL2+/TNFa-/IFNg-, Day 37 | 28 [4 to 49] | 4 [4 to 4] | 4 [4 to 6] | 4 [4 to 4] | 4 [4 to 18] | 4 [4 to 28]
  CD40L-/IL2+/TNFa-/IFNg-, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L-/IL2+/TNFa-/IFNg-, Day 60 | 4 [4 to 15.5] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 20] | 4 [4 to 19]
  CD40L-/IL2+/TNFa-/IFNg-, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L-/IL2+/TNFa-/IFNg-, Day 210 | 4 [4 to 13] | 38 [4 to 98] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 19]

25. Secondary Outcome: Frequency of CD8+ T-cells M72-specific Expressing Cytokines in Any Combination
Description: as for outcome 9
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD8+ T-cells/million cells
  CD40L-/IL2-/TNFa+/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L-/IL2-/TNFa+/IFNg+, Day 0 | 4 [4 to 199.5] | 4 [4 to 73] | 4 [4 to 47] | 30 [4 to 286] | 4 [4 to 37] | 4 [4 to 45]
  CD40L-/IL2-/TNFa+/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L-/IL2-/TNFa+/IFNg+, Day 7 | 50 [30.5 to 101] | 4 [4 to 5] | 32 [4 to 109] | 4 [4 to 284] | 4 [4 to 104] | 9 [4 to 102]
  CD40L-/IL2-/TNFa+/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L-/IL2-/TNFa+/IFNg+, Day 30 | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 107] | 91.5 [4 to 1024] | 4 [4 to 39] | 4 [4 to 73]
  CD40L-/IL2-/TNFa+/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L-/IL2-/TNFa+/IFNg+, Day 37 | 41 [4 to 66] | 4 [4 to 53] | 28.5 [4 to 285] | 28 [4 to 228] | 4 [4 to 30] | 4 [4 to 85]
  CD40L-/IL2-/TNFa+/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L-/IL2-/TNFa+/IFNg+, Day 60 | 19 [4 to 144] | 35 [4 to 66] | 29 [4 to 149] | 58 [4 to 432] | 4 [4 to 39] | 4 [4 to 45]
  CD40L-/IL2-/TNFa+/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L-/IL2-/TNFa+/IFNg+, Day 210 | 51 [4 to 264] | 4 [4 to 4] | 4 [4 to 184] | 4 [4 to 101] | 4 [4 to 27] | 4 [4 to 30.5]
  CD40L-/IL2-/TNFa+/IFNg-, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L-/IL2-/TNFa+/IFNg-, Day 0 | 21 [4 to 80] | 4 [4 to 61] | 4 [4 to 36] | 7.5 [4 to 37] | 25.5 [4 to 57] | 4 [4 to 18]
  CD40L-/IL2-/TNFa+/IFNg-, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L-/IL2-/TNFa+/IFNg-, Day 7 | 17 [4 to 61] | 4 [4 to 5] | 4 [4 to 59] | 4 [4 to 82] | 20.5 [4 to 39] | 4 [4 to 27]
  CD40L-/IL2-/TNFa+/IFNg-, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L-/IL2-/TNFa+/IFNg-, Day 30 | 4 [4 to 4] | 80 [4 to 156] | 4 [4 to 67.5] | 47.5 [6 to 123] | 20.5 [4 to 67] | 24.5 [4 to 71]
  CD40L-/IL2-/TNFa+/IFNg-, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L-/IL2-/TNFa+/IFNg-, Day 37 | 40 [4 to 128] | 4 [4 to 69] | 36.5 [4 to 112] | 4 [4 to 43] | 4 [4 to 27] | 5 [4 to 64]
  CD40L-/IL2-/TNFa+/IFNg-, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L-/IL2-/TNFa+/IFNg-, Day 60 | 16 [4 to 54] | 4 [4 to 4] | 4 [4 to 89] | 18.5 [4 to 90] | 20 [4 to 56] | 4.5 [4 to 30]
  CD40L-/IL2-/TNFa+/IFNg-, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L-/IL2-/TNFa+/IFNg-, Day 210 | 4 [4 to 4] | 4 [4 to 8] | 4 [4 to 4] | 4 [4 to 42] | 4 [4 to 60] | 4 [4 to 29]

26. Secondary Outcome: Frequency of CD8+ T-cells M72-specific Expressing Immune Markers in Any Combination
Description: as for outcome 7
Time Frame: Prior to dose 1 (Day 0), post-dose 1 (Days 7 and 30), post-dose 2 (Days 37, 60 and 210)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: CD8+ T-cells/million cells
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
Number analyzed (Participants) | 6 | 3 | 18 | 22 | 37 | 36
CD8+ T-cells/million cells
  CD40L-/IL2-/TNFa-/IFNg+, Day 0: number analyzed (Participants) | 4 | 3 | 15 | 22 | 30 | 30
  CD40L-/IL2-/TNFa-/IFNg+, Day 0 | 54.5 [25.5 to 821] | 6 [4 to 95] | 70 [12 to 541] | 216.5 [57 to 1831] | 54.5 [4 to 159] | 78.5 [25 to 349]
  CD40L-/IL2-/TNFa-/IFNg+, Day 7: number analyzed (Participants) | 4 | 3 | 13 | 15 | 26 | 28
  CD40L-/IL2-/TNFa-/IFNg+, Day 7 | 89 [36.5 to 893.5] | 9 [4 to 31] | 152 [4 to 575] | 205 [90 to 1660] | 69.5 [43 to 830] | 90.5 [4.5 to 484.5]
  CD40L-/IL2-/TNFa-/IFNg+, Day 30: number analyzed (Participants) | 5 | 2 | 16 | 16 | 34 | 34
  CD40L-/IL2-/TNFa-/IFNg+, Day 30 | 96 [26 to 163] | 118 [4 to 232] | 127.5 [13 to 327.5] | 386.5 [27 to 1969.5] | 64.5 [4 to 438] | 151.5 [28 to 467]
  CD40L-/IL2-/TNFa-/IFNg+, Day 37: number analyzed (Participants) | 5 | 3 | 18 | 19 | 34 | 34
  CD40L-/IL2-/TNFa-/IFNg+, Day 37 | 48 [4 to 78] | 33 [4 to 81] | 100.5 [48 to 326] | 229 [4 to 1022] | 46.5 [4 to 179] | 83.5 [4 to 335]
  CD40L-/IL2-/TNFa-/IFNg+, Day 60: number analyzed (Participants) | 4 | 2 | 15 | 18 | 31 | 32
  CD40L-/IL2-/TNFa-/IFNg+, Day 60 | 147.5 [55 to 824.5] | 4 [4 to 4] | 70 [4 to 1116] | 172 [18 to 1492] | 13 [4 to 65] | 59 [4 to 310]
  CD40L-/IL2-/TNFa-/IFNg+, Day 210: number analyzed (Participants) | 6 | 3 | 13 | 17 | 37 | 36
  CD40L-/IL2-/TNFa-/IFNg+, Day 210 | 286.5 [48 to 469] | 4 [4 to 59] | 51 [4 to 245] | 85 [4 to 628] | 69 [4 to 233] | 60 [22 to 232.5]

ADVERSE EVENTS:
Time Frame: Solicited AEs: during the 7-day (Days 0-6) post-vaccination period; Unsolicited AEs: during the 30-day (Days 0-29) post-vaccination period; SAEs: up to Day 210.
Description: Results presented per group consist of a summary of the events (SAEs and AEs other than SAEs, respectively) reported, compiling overall number of subjects with events across the different periods of assessment.
Arm/Group | TB Treatment GSK 692342 Group | TB Treatment Saline Group | TB Treated GSK 692342 Group | TB Treated Saline Group | TB Naive GSK 692342 Group | TB Naive Saline Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/24 | 0/25 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 2/24 | 2/25 | 1/40 | 0/40
Other Adverse Events (participants affected / at risk) | 6/7 | 3/6 | 24/24 | 14/25 | 40/40 | 26/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TB Treatment GSK 692342 Group (N=7) | TB Treatment Saline Group (N=6) | TB Treated GSK 692342 Group (N=24) | TB Treated Saline Group (N=25) | TB Naive GSK 692342 Group (N=40) | TB Naive Saline Group (N=40)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TB Treatment GSK 692342 Group (N=7) | TB Treatment Saline Group (N=6) | TB Treated GSK 692342 Group (N=24) | TB Treated Saline Group (N=25) | TB Naive GSK 692342 Group (N=40) | TB Naive Saline Group (N=40)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 1 (1) | 18 (24) | 4 (6) | 25 (32) | 6 (8)
Pain (General disorders) | 6 (11) | 1 (2) | 22 (41) | 3 (3) | 39 (74) | 8 (11)
Swelling (General disorders) | 5 (8) | 0 (0) | 12 (19) | 3 (3) | 22 (29) | 2 (2)
Fatigue (General disorders) | 3 (4) | 2 (3) | 17 (27) | 8 (11) | 36 (52) | 10 (15)
Gastrointestinal symptoms (Gastrointestinal disorders) | 2 (2) | 0 (0) | 10 (11) | 4 (5) | 16 (18) | 6 (8)
Malaise (General disorders) | 3 (4) | 2 (3) | 16 (22) | 6 (7) | 35 (46) | 9 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 18 (27) | 5 (8) | 34 (52) | 7 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 4 (4) | 3 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 5 (9) | 2 (2) | 16 (22) | 6 (6) | 25 (36) | 12 (18)
Pyrexia (General disorders) | 4 (4) | 1 (1) | 11 (11) | 0 (0) | 17 (18) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to a safety signal found at a planned interim safety review, further conduct of this safety study is not recommended hence the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.